CLINICAL TRIAL: NCT04026659
Title: The Feasibility of Implementing an Exercise Programme for Deconditioned Cancer Survivors in a National Cancer Centre: FIXCAS Study
Brief Title: The Feasibility of Implementing an Exercise Programme for Deconditioned Cancer Survivors
Acronym: FIXCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Irish Cancer Society (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Grainne Sheill, Principal Investigator, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STS19SHE
Record Dates: First submitted 2019-07-02; First posted 2019-07-19 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Cancer
Keywords: Exercise; Rehabilitation
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-modal exercise programme (Experimental): The 10-week multi-modal exercise programme will comprise of twice weekly supervised group-based exercise sessions. Each exercise session will last approximately 1 hour and consist of a combination of aerobic, resistance and balance and flexibility exercises.
  Interventions: Other: Multi-modal exercise

INTERVENTIONS:
Other: Multi-modal exercise — A combination of aerobic, resistance, balance and flexibility exercises will be included. Aerobic exercise will consist of 20 to 30 min of moderate intensity exercise using a variety of modalities. Heart rate will be monitored using Polar hear rate monitors (target intensity 40-70% heart rate reserve) and the BORG Rating of Perceived Exertion (12-15). Resistance exercise will target the large muscle groups of the upper and lower extremities, be performed at 40% to 70% of the one repetition maximum (1-RM) and consist of two sets of 10-15 repetitions. Flexibility and balance exercise will also be included in the twice weekly programme. A home exercise programme will encourage participants to be moderately physically active for at least 30 minutes, three times per week in addition to the supervised programme.

SUMMARY:
As both the number of cancer survivors and the length of survival time are increasing, long-term health issues related to cancer and its treatment are becoming more prevalent. Research suggests that exercise can mitigate a number of negative health consequences in cancer survivors and improve physical function and quality of life. Multi-modal exercise interventions have been proposed as a cornerstone for survivorship care. However, studies evaluating exercise programmes within the Irish population are lacking. The aim of the study is to evaluate the introduction, implementation and acceptability of a multi-modal exercise rehabilitation programme for deconditioned cancer survivors in a real-world, standard practice setting.

DETAILED DESCRIPTION:
There are currently more than 150,000 cancer survivors in Ireland, and this number continues to rise. Subsequently, as both the number of cancer survivors and the length of survival time are increasing, long-term health issues related to cancer and its treatment are becoming more prevalent.

Depending on the specific treatment exposures, cancer survivors can face numerous adverse consequences of cancer treatment. Numerous systematic reviews demonstrate that exercise can mitigate a number of these factors in cancer survivors and improve quality of life, cardiorespiratory fitness, physical functioning, fatigue and can optimise functional status, preserving the ability to remain in the workforce and fulfil other life roles.

Despite the robust body of existing literature, addressing the long term side effects of cancer is a major challenge for health care policy and the integration and delivery of exercise rehabilitation and survivorship into standard clinical cancer care in Ireland continues to remain the exception rather than the norm. Internationally, models of cancer survivorship care have been developing rapidly in recent years, many centring on the provision of exercise rehabilitation programmes across diverse delivery settings. However, referral to exercise specialists is not a part of the standard care received by oncology patients in Ireland with a distinct lack of rehabilitation services available for cancer survivors.

The aim of the FIXCAS study is to examine the feasibility of implementing a 10 week multi-modal exercise rehabilitation programme to deconditioned cancer survivors in a National Cancer Centre.

This single-arm prospective feasibility study will evaluate the introduction, implementation and acceptability of an exercise rehabilitation programme for deconditioned cancer survivors in a real-world, standard practice setting. A convenience sample of cancer survivors (n=40) aged 18 or older that have completed treatment with curative intent attending outpatient oncology services in a National Cancer Centre will be recruited. Participants will undergo a 10-week multi-modal exercise programme. Feasibility will be evaluated in terms of recruitment, adherence and compliance to the programme. Secondary outcomes will examine physical function and quality of life measures. In addition, the acceptability of the programme will be assessed through patient feedback.

The study results will be used to optimise the intervention content, and may serve as the foundation for a larger definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Diagnosis of solid tumour
* Completion of chemotherapy and/or radiotherapy with curative intent within the preceding 2-6 months
* Medically fit to participate in moderate physical activity

Exclusion Criteria:

* Moderate or severe cognitive impairment
* Current pregnancy
* Individuals receiving treatment in the palliative setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Programme feasibility - recruitment rates as assessed by percentage of eligible study population that consent to participation | 24 weeks
  The primary outcome of this study will be its feasibility aspects including recruitment rates (percentage of eligible study population that consent to participation)
Programme feasibility - adherence as assessed by the number of prescribed supervised and unsupervised sessions completed by participants | 24 weeks
  The primary outcome of this study will be its feasibility aspects including programme adherence (number of prescribed supervised and unsupervised sessions completed by participants)
Programme feasibility - retention rates as assessed by the number of participants completing the programme and number of dropouts | 24 weeks
  The primary outcome of this study will be its feasibility aspects including programme retention rates (number of participants completing the programme and number of dropouts)
Programme feasibility - acceptability of the intervention as assessed by qualitative interviews | 24 weeks
  Acceptability of the intervention will be explored through qualitative interviews. Key stakeholders, namely participants in the exercise intervention and health professionals referring to the exercise programme will be invited to participate in semi-structured interviews. Health professionals (n=8-10) referring to the programme will be interviewed to examine their experience of referring to the FIXCAS programme to identify barriers and facilitators to referral and to determine areas for review and further development. Patients (n=10-15) will be asked to evaluate satisfaction with the intervention. Open-ended questions will be used to encourage reflection and elaboration on different aspects of the programme. The interviews will be recorded and transcribed, and data analysis of the interviews will occur through content analysis using simple descriptive thematic analyses.

SECONDARY OUTCOMES:
Change in physical fitness | Baseline and 10 weeks
  Physical fitness will be measured by the 6 minute walk test (6MWT), a valid and reliable measure of physical fitness in people with cancer which will be performed according to the American Thoracic Society (ATS) Guidelines.
Change in physical activity | Baseline and 10 weeks
  Self-reported physical activity will be collected using the International Physical Activity Questionnaire (IPAQ). The IPAQ is a self-report measure of physical activity on a 12-item scale. The total score will be summed within each physical activity domain to estimate the total time spent in occupational, transport, household, and leisure related physical activity, as well as total time reported sitting per week. The total score ranges from 0 to the highest number of time (hours) that the participants can spent on physical activity. A higher score means higher level of physical activity.
Change in physical performance | Baseline and 10 weeks
  Physical performance will be measured by a Short Physical Performance Battery (SPPB). The SPPB is a simple test of standing balance, usual walking speed (4-metre gait speed) and ability to stand from a chair, which reflects global physical functioning and frailty. Each section is scored between 0 (worst) - 4 (best) and the total score ranges from 0 (worst performance) to 12 (best performance).
Change in lower limb strength | Baseline and 10 weeks
  Leg extension 1 repetition maximum will be measured.
Change in Quality of Life (QoL) as assessed by the European Organisation for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30) | Baseline, 10 weeks, 24 weeks
  Quality of life is evaluated through the internationally established EORTC-QLQ-C30. The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms.
  All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Change in Quality of Life (QoL) as assessed by the Euro-QoL-5 Dimension-5 Level (EQ-5D-5L). | Baseline, 10 weeks, 24 weeks
  EQ-5D-5L is a generic quality of life measure. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the visual analogue scale (VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to choose one of 5 levels that best describes their health on that day: "no problem" (1), "slight" (2), "moderate" (3), "severe" (4), or "unable/extreme" (5). The VAS is the participant's rating of their health on a scale of 0 "worst health you can imagine" to 100 "best health you can imagine".
Change in fatigue | Baseline and 10 weeks
  Fatigue will be assessed using the Brief Fatigue Inventory (BFI).The BFI is a 9-item, 11-point rating scale developed to assess subjective fatigue. The first three questions measure fatigue severity from 0, indicating "no fatigue," to 10, indicating "as bad as you can imagine," at current, usual, and worst levels. The following six questions assess fatigue interference with daily activities including general activity, mood, walking ability, normal work (both inside and outside the home), relations with other people, and enjoyment of life. Response options range from 0, indicating "does not interfere," to 10, indicating, "completely interferes." Higher scores on the BFI correspond to greater self-reported levels of fatigue.
Change in incontinence (prostate cancer only) | Baseline and 10 weeks
  Prostate cancer survivors will complete the International Consultation on Incontinence Questionnaire (ICIQ). The ICIQ is a self-reported survey and screening tool for incontinence and asks for rating of symptoms in the past 4 weeks. The sum score of items 3, 4, 5 is calculated for the actual score. Change in mean test scores range = 0 - 21; low score = mild symptoms, high score = significant impact on quality of life.
Change in sexual function (prostate cancer only) | Baseline and 10 weeks
  Prostate cancer survivors will complete the Brief Male Sexual Function Inventory (BSFI). The questions in the BSFI are evaluated on a series of 5-item Likert scales, from 0 or 1 points to 4 or 5 points. Scores are calculated for each of the 5 functional domains, along with a total BSFI score. Whilst there is no specific cut-off, the closer the score is to 1, the higher the lower urinary tract symptom severity and impairment to sexual function. Scores closer to 45 are considered to indicate less severe symptoms and little to no sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Sheill, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- St. James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devenney K, Murphy N, Ryan R, Grant C, Kennedy J, Manecksha RP, Sheils O, McNeely ML, Hussey J, Sheill G. The feasibility of implementing an exercise programme for deconditioned cancer survivors in a national cancer centre: FIXCAS Study. HRB Open Res. 2020 Dec 18;2:24. doi: 10.12688/hrbopenres.12925.2. eCollection 2019. PMID 33870087